CLINICAL TRIAL: NCT03135379
Title: Comparison of Patient Satisfaction Using Heated Versus Room Temperature Ultrasound Gel: a Single-blind Randomized Controlled Trial
Brief Title: Comparison of Patient Satisfaction Using Heated Versus Room Temperature Ultrasound Gel
Acronym: HUGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Program Director for Research, Emergency Medicine, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: C.2016.046d
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Ultrasound

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A heat-resistant glove, ULine Terry Cloth Glove (Appendix F), will be used by the investigators to handle the ultrasound gels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heated gel (Experimental): Patient undergoes ultrasound study using the intervention of heated ultrasound gel.
  Interventions: Device: Heated ultrasound gel
- Room temperature gel (Placebo Comparator): Patient undergoes ultrasound study using the intervention of room temperature gel.
  Interventions: Device: Room temperature gel

INTERVENTIONS:
Device: Heated ultrasound gel — Gel stored in Thermasonic Gel Warmer (Model 82-03 LED, 120V) set to "medium" setting (102 degree fahrenheit).
  Arms: Heated gel
Device: Room temperature gel — Gel stored in Thermasonic Gel Warmer (Model 82-03 LED, 120V) turned off.
  Arms: Room temperature gel

SUMMARY:
The purpose of this single-blind, randomized control trial will be to investigate whether simply having warmed gel, as compared to room-temperature gel, during a bedside ultrasound significantly improves patient satisfaction scores.

DETAILED DESCRIPTION:
ED physicians who identify that a patient will require an ultrasound will page the ultrasound team as part of standard of care. At that time, an investigator will obtain verbal consent from the patient and provide an information sheet to help explain study details/answer any questions. The patient will then be randomized to either warmed gel or room temperature gel. Investigators will handle the gel using a heat-resistant glove (ULine Terry Cloth Glove) to maintain blinding to the gel temperature. A bedside ultrasound study will then be performed by emergency physicians not otherwise involved in the study using the study gel. Immediately upon ultrasound completion, the patients will complete a satisfaction survey. The images from the study will be saved and subsequently reviewed by an emergency physician with fellowship training in ultrasound to score image quality from 1 (low) to 5 (high).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-89 years
* Patients require bedside ultrasound

Exclusion Criteria:

* Patients under age 18
* Patients over age 89
* Pregnant women
* Altered mental status
* Incarcerated
* Military basic trainees
* Primary language other than English
* Patients with open or broken skin over areas requiring ultrasound gel application

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Krainin, MD, Principal Investigator — benjamin.m.krainin.mil@mail.mil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cydulka RK, Tamayo-Sarver J, Gage A, Bagnoli D. Association of patient satisfaction with complaints and risk management among emergency physicians. J Emerg Med. 2011 Oct;41(4):405-11. doi: 10.1016/j.jemermed.2010.10.021. Epub 2011 Jan 7. PMID 21215554
- [Background] Levin DC, Rao VM, Parker L, Frangos AJ. Continued growth in emergency department imaging is bucking the overall trends. J Am Coll Radiol. 2014 Nov;11(11):1044-7. doi: 10.1016/j.jacr.2014.07.008. Epub 2014 Nov 3. PMID 25439619
- [Background] Singer AJ, Thode HC Jr. Determination of the minimal clinically significant difference on a patient visual analog satisfaction scale. Acad Emerg Med. 1998 Oct;5(10):1007-11. doi: 10.1111/j.1553-2712.1998.tb02781.x. PMID 9862594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heated Gel | Room Temperature Gel
Started | 62 | 62
Completed | 61 | 59
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heated Gel | Room Temperature Gel | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (17.6) | 42.0 (18.5) | 41.7 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 32 | 51
  Male | 42 | 27 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Measured on 100-mm visual analogue scale. This scale is a horizontal line on a sheet of paper measuring 100 mm. The scale ranges from 0 on the left (representing "completely unsatisfied") to 100 on the right (representing "completely satisfied"). We instructed subjects to draw a single vertical mark through the horizontal line to represent how satisfied they were with their overall emergency department visit.
Time Frame: Immediately upon completion of ultrasound examination
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Heated Gel | Room Temperature Gel
Number analyzed (Participants) | 61 | 59
units on a scale | 87.6 [84.8 to 90.1] | 83.9 [79.4 to 87.6]

2. Secondary Outcome: Ultrasound Image Quality
Description: Measured 1 (low) to 5 (high) by an attending emergency physician who has completed ultrasound fellowship.
Time Frame: Within 1 week of completion of ultrasound examination
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Heated Gel | Room Temperature Gel
Number analyzed (Participants) | 40 | 39
units on a scale | 4 [3 to 4] | 4 [4 to 4]

ADVERSE EVENTS:
Time Frame: 30 minutes
Arm/Group | Heated Gel | Room Temperature Gel
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03135379/Prot_SAP_000.pdf